CLINICAL TRIAL: NCT00430274
Title: Photographic Imaging of the Retina and Optic Nerve Head of Glaucoma Patients and Normal Controls
Status: Completed | Type: Observational
Sponsor: Selim Orguel (Other)
Responsible Party: Sponsor-Investigator, Selim Orguel, Prof. Dr., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 073-GRM-2006-001
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma
Keywords: glaucoma; retinal gliosis-like alterations; optical coherence tomography; automated microperimetry
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retinal structures are difficult to visualize because the retina is optically transparent. In glaucoma, the microglia in the retina becomes activated in eyes with glaucomatous damage. The microglia forms a dense meshwork which resembles gliosis-like alterations, which may increase light scattering. With appropriate technology, increased reflection and light scattering from the retina may be detected in eyes of glaucoma patients.

In this study, we investigate whether clinically observable retinal gliosis-like alterations occur more often in patients with glaucoma than in non-glaucomatous controls, and whether gliosis-like alterations are associated with a vasospastic propensity.

DETAILED DESCRIPTION:
Glaucoma is an optic neuropathy characterized by a progressive loss of retinal ganglion cells and cupping of the optic nerve head associated with visual function defects. Increased intraocular pressure and vascular alterations such as unsteady blood flow have been implicated in the pathogenesis of glaucoma. While glaucoma changes occur in both the retina and the optic nerve head, clinical diagnosis normally focuses on optic nerve head. However, histomorphologic and immunohistochemistry studies have shown that glial cells in the retina (astrocytes and Müller cells) are also activated in glaucoma. In addition, some patients with glaucoma have clinically patchy alteration in the retina resembling epiretinal gliosis but without visual disturbance, thus the term "gliosis-like alterations" was used previously. At present however, it is unknown whether gliosis-like alterations are associated with a specific type of glaucoma (i.e. high- or normal-tension glaucoma) or with vascular dysregulation. Moreover, it remains unclear whether gliosis-like alterations may also occur in the elderly patients without glaucoma as an aging process of the retina. Retinal structures are difficult to visualize and details difficult to be imaged on a photograph because the retina is optically transparent. Blue light scatters more than red light. This is the reason why the retinal nerve fiber layer can to some extent be better visualized with red-free light. The extensions of the astrocytes in the retina form a fine meshwork, which becomes denser and irregular as these astrocytes are activated. The size and numbers of glial cells increase, as the neural cell damage advances. These changes, in turn, may increase the light scattering. With appropriate technology, increased reflection and light scattering from the retina may be detected in the retina of glaucoma patients. The purpose of the study is to evaluate whether gliosis-like alterations do occur more often in glaucoma.

The retina of patients and healthy controls alike will be photographically documented with a digital fundus camera as well as with optical coherence tomography and automated microperimetry that enables to correlate objectively local morphologic aspects and changes of the retina with local functional measurements. Possible causes for secondary retinal gliosis will be excluded in a thorough clinical examination including slit-lamp examination and dilated direct fundoscopy. The examination techniques and interventions used in this study are routine clinical practice and do not expose patients or controls to undue risk.

ELIGIBILITY:
Inclusion Criteria:

For NTG patients :

* untreated intraocular pressure equal to or less than 21mmHg or
* median intraocular pressure equal to or less than 20mmHg

For HTG patients:

* mean untreated intraocular pressure more than 21mmHg

For both:

* open drainage angles on gonioscopy
* typical optic disc damage with glaucomatous cupping and thinning of neuroretinal rim
* absence of any secondary cause for a glaucomatous optic neuropathy
* visual field defects congruent to glaucomatous disc damage (disc/field correlation)

Healthy subjects:

* no history of ocular diseases
* no current topical medication
* no drug or alcohol abuse
* best corrected visual acuity above 20/25 in both eyes
* no pathological findings upon a slit-lamp examination and fundoscopy
* IOP < 21 mmHg in both eyes

Exclusion Criteria:

For NTG and HTG patients:

* any other form of retinal or neuroophthalmological disease that could cause gliosis-like retinal alterations or result in visual field defects
* history of chronic or recurrent severe inflammatory eye disease
* history of ocular trauma or intraocular surgery
* history of infection or inflammation within the past 3 months
* history and clinical evidence for other retinal disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with vascular dysregulation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Eye Clinic, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No